Date: March 2015

Results of RBM device testing of newborn baby temperature measurement in different temperature ranges and in different settings of St John's Medical College Hospital, Bangalore (2015)

(a) Normal temperature range (above 35.5°C) in neonatal ICU setting

| Experiment date | Newborn<br>SI No. | No of temp readings | Temp_device (Tdev) | Temp_probe<br>(Tp) | Tdev-Tp<br>diff |
|---|---|---|---|---|---|
| 09-02-2015 | 1 | 12 | 36.62 | 36.57 | 0.05 |
| 11-02-2015 | 2 | 12 | 35.78 | 36.56 | -0.78 |
| 12-02-2015 | 3 | 12 | 35.66 | 36.34 | -0.68 |
| 18-02-2015 | 4 | 12 | 36.24 | 36.64 | -0.4 |
| Average | | | 36.08 | 36.53 | -0.45 |

Average 36.08 36.53 -0.45

(b) Temperature range around 33°C for a baby undergoing therapeutic cooling for birth asphyxia in neonatal ICU setting

| Experiment date | Newborn<br>SI No. | • | Temp_device (Tdev) | Temp_probe (Tp) | Tdev-Tp<br>diff |
|---|---|---|---|---|---|
| 25-03-2015 | 5 | 12 | 33.10 | 33.15 | 0.05 |

(c) Temperature range around 34°C for a baby undergoing re-warming after therapeutic cooling for birth asphyxia in neonatal ICU setting

| Experiment date | Newborn<br>SI No. | No of temp readings | Temp_device (Tdev) | Temp_probe<br>(Tp) | Tdev-Tp<br>diff |
|---|---|---|---|---|---|
| 27-03-2015 | 5 | 12 | 33.95 | 33.92 | 0.03 |

Temp\_device (Tdev) = temperature acc to RBM device

Temp\_probe (Tp) = temperature acc to the NICU radiant warmer probe

Tdev-Tp diff = difference in temperature b/n the two thermometers (values >0.5° difference marked in red)

(d) Temperature readings in the early morning time (b/n 4.00 to 5.00 a:m) for a well-baby in the postnatal ward with mother

| Experiment date | Newborn<br>SI No. | No of temp readings | Temp_device (Tdev) | Temp_digital<br>(Tdig) | Tdev-Tdig<br>diff |
|---|---|---|---|---|---|
| 26-03-2015 | 1 | 12 | 36.61 | 36.61 | 0.00 |
| 27-03-2015 | 2 | 12 | 37.00 | 36.82 | 0.18 |
| 27-03-2015 | 3 | 12 | 37.00 | 36.79 | 0.21 |
| | | | 22.2= | 20 = 4 | 0.10 |

Average 36.87 36.74 0.13